CLINICAL TRIAL: NCT02889406
Title: Clinical and Metabolic Efficacy of the Motivational Approach, Coordinated Between Primary Care and the Clinical Health Services for Childhood Obesity Treatment: Randomized Clinical Trial
Brief Title: Motivation Approach for Childhood Obesity Treatment
Acronym: OBEMAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/01411
Record Dates: First submitted 2016-07-11; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational intervention (Experimental): Following the motivational interviewing schema, structured in 2 phases of treatment (motivational and intervention) and organised in 11 visits (one each month). The first and last visits will be performed in consultations of endocrinology unit from referral hospitals; the other visits will be held in paediatric primary care setting. Visits will be scheduled monthly and each one will last between 15 and 20 minutes.
  In addition to individualized visits, three group workshops focused in nutrition education for families will be organized. Each workshop will last 45 minutes and will target parents/mothers and obese children, separately.
  Interventions: Behavioral: Motivational intervention
- Control group (No Intervention): Children who are assigned to the control group will follow the usual treatment performed in paediatrics, what is following the Clinical Practice Guideline on the prevention and treatment of child and adolescent obesity. Monthly visits will be conducted in which weight, height and waist circumference will be measured and compliance with the initial advice will be reviewed.

INTERVENTIONS:
Behavioral: Motivational intervention — motivational interviewing schema
  Arms: Motivational intervention

SUMMARY:
In a recent study, we have demonstrated that the motivational therapy approach to treat childhood obesity is highly effective at clinical and metabolic levels. This efficacy has been proved in a clinical outpatient setting. However, a standardized collaborative approach between the clinic and the primary care services would allow a faster and easier approach to childhood obesity treatment. Furthermore, this motivational and educational intervention would benefit from the current technologic facilities, the long term effect of the education at group level, in terms of food shopping plan, healthy, fast and cheap cooking methods that would be useful specially in low income families (with a higher prevalence of childhood obesity).

The aim of this study is assessing the clinical and metabolic efficacy of a family intervention, coordinated between the clinical and primary care services from the Tarragona health-care region, using a motivational therapy at individual and group levels, which involves e-Health tools (wearable), focusing on families with an 8 to 13 years old obese child.

The design will be a clustered randomized control trial, with an intervention group that will receive a multicomponent motivational and educational plan which will be compared to a control group receiving the usual recommendations performed in primary care centres (n=167 per group). The treatment of both study groups will last 12 months and will be performed at the primary care centres. In parallel, the study team will validate the methodology used to assess body composition in obese children as well as the changes produced by the intervention.

DETAILED DESCRIPTION:
MAIN OBJECTIVE To evaluate the effectiveness of a motivational intervention for the treatment of childhood obesity, coordinated between primary care and specialized services, multicomponent, integrating techniques of fast and healthy cooking and eHealth tools (wearable), compared to the usual intervention performed in paediatrics.

SPECIFIC OBJECTIVES

1. To evaluate the effectiveness of a multicomponent motivational intervention compared to usual intervention performed in regular paediatrics clinical practice

   1. On BMI control of obese children between 8 and 13 years old
   2. On metabolic control of obese children between 8 and 13 years old,
   3. On increasing physical activity of obese children between 8 and 13 years old,
   4. On acquiring a healthy eating pattern in obese children between 8 and 13 years old.
2. To establish methodological background for implantation of a motivational intervention coordinated between primary care services and specialized services.
3. To validate the use of bioelectrical impedance analysis (BIA) and dual X-ray absorptiometry (DXA) in the follow up and treatment of childhood obesity compared to four-compartment model of body composition.

5. METHODOLOGY

5.1 Design Randomized controlled clinical trial cluster, with an intervention group (IG) which will receive 12 months of motivational counselling, together with workshops focused on family nutrition education and techniques of fast and healthy cooking and physical activity; and with eHealth tools (wearable) to support; and a control group (CG) that will follow the usual recommendations.

5.2 STUDY POPULATION The Health Region of Tarragona includes a population of 600,000 people (36,000 children from 8 to 13 years). With regard to the 6.6% of childhood obesity prevalence in our country (Schroder 2014), we estimate an eligible population of 2376 obese children aged 8-13 years old.

5.3 SAMPLE SIZE The number of individuals of a simple random design, multiplied by the design effect has been considered to calculate the sample size of each stratum (Basic Care Unit). Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 98 subjects were needed in each group to detect a difference equal to or greater than 0.36 units of BMI z-score. It is assumed that common standard deviation is 0.75. A 30% lost to follow up rate (GRANMO 7.12) has been estimated. To calculate the design effect, estimates of intracluster correlation coefficient in cluster randomized trials in primary care are generally lower than 0.05. The effect of the design corresponds to 1.7. Assuming these values, the final size of the study sample would be of 167 subjects in each group (12 individuals for each primary care centre, in 15 basic care units (BCUs)).

5.4 RANDOMIZATION AND BLINDING Basic Care Units (BCU) doctor-nurse are the unit of randomization. Randomization will be 1: 1 and will be made with EPIDAT 3.0 statistical program. Given the nature of the intervention participants or researchers cannot be blinded. Professional in charge of statistical analysis will be blinded as well.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients which are between 8 and 13 years at enrolment, using as diagnostic criteria of obesity values of body mass index (BMI) above the 97th percentile of Hernandez references from 1988

Exclusion Criteria:

* Participants who do not sign the informed consent
* Children with eating disorders
* Families not available to attend to intervention scheduled visits
* Simultaneous participation in another randomized trial
* Presence of endocrine disorders (GH disorder, hypothyroidism, Cushing's disease, precocious puberty or other)
* Illiteracy or lack knowledge of local languages

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 334 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI z-score | 12 months
  Changes in BMI z-score between the first visit and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Josep Basora, MD, Study Director — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Unitat Suport a la Recerca (Tarragona-Reus) Idiap Jordi Gol, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luque V, Feliu A, Escribano J, Ferre N, Flores G, Monne R, Gutierrez-Marin D, Guillen N, Munoz-Hernando J, Zaragoza-Jordana M, Gispert-Llaurado M, Rubio-Torrents C, Nunez-Roig M, Alcazar M, Ferre R, Basora JM, Hsu P, Alegret-Basora C, Arasa F, Venables M, Singh P, Closa-Monasterolo R. The Obemat2.0 Study: A Clinical Trial of a Motivational Intervention for Childhood Obesity Treatment. Nutrients. 2019 Feb 16;11(2):419. doi: 10.3390/nu11020419. PMID 30781525